CLINICAL TRIAL: NCT04761081
Title: Is Physical Activity Associated With the Tethering and Migration of Pro-inflammatory Monocytes in White European and South Asian Males With and Without Central Obesity.
Brief Title: Is Physical Activity, Obesity, and Ethnicity Associated With the Tethering and Migration of Pro-inflammatory Monocytes?
Status: Completed | Type: Observational
Sponsor: Loughborough University (Other)
Responsible Party: Principal Investigator, Nicolette Bishop, Professor, Loughborough University
Other Study IDs: 2020-1885-2140
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Physical Activity; Central Obesity; Inflammation
Keywords: Physical activity; Central obesity; Ethnicity; Inflammation
MeSH Terms: conditions — Motor Activity; Obesity, Abdominal; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma samples will be stored for the measurement of metabolic markers (triacylglycerol, glucose, total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, non-esterified free fatty acids, c-reactive protein, interleukin-6.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- South Asians who are lean: The south Asian group who are lean will be of south Asian ethnicity and a waist circumference <90cm.
  The group will receive an accelerometer (Actigraph GT3x) to wear for 7 days to measure habitual physical activity. They will then provide a single blood donation in a fasted state which we will use to quantify the migration of pro-inflammatory monocytes towards adipose tissue specific media. This will then be compared to the other 3 groups to investigate the interaction between ethnicity, central obesity, and physical activity with the migration of pro-inflammatory monocytes.
  Metabolic markers will be analysed and presented in a participant characteristics table.
  Interventions: Behavioral: Habitual physical activity assessment
- South Asians with central obesity: The south Asian group with central obesity will be of south Asian ethnicity and a waist circumference of 90cm or greater.
  The group will receive an accelerometer (Actigraph GT3x) to wear for 7 days to measure habitual physical activity. They will then provide a single blood donation in a fasted state which we will use to quantify the migration of pro-inflammatory monocytes towards adipose tissue specific media. This will then be compared to the other 3 groups to investigate the interaction between ethnicity, central obesity, and physical activity with the migration of pro-inflammatory monocytes.
  Metabolic markers will be analysed and presented in a participant characteristics table.
  Interventions: Behavioral: Habitual physical activity assessment
- White Europeans who are lean: The white European group who are lean will be of white European ethnicity and a waist circumference <94cm.
  The group will receive an accelerometer (Actigraph GT3x) to wear for 7 days to measure habitual physical activity. They will then provide a single blood donation in a fasted state which we will use to quantify the migration of pro-inflammatory monocytes towards adipose tissue specific media. This will then be compared to the other 3 groups to investigate the interaction between ethnicity, central obesity, and physical activity with the migration of pro-inflammatory monocytes.
  Metabolic markers will be analysed and presented in a participant characteristics table.
  Interventions: Behavioral: Habitual physical activity assessment
- White Europeans with central obesity: The white European group with central obesity will be of white European ethnicity and a waist circumference of 94cm or greater.
  The group will receive an accelerometer (Actigraph GT3x) to wear for 7 days to measure habitual physical activity. They will then provide a single blood donation in a fasted state which we will use to quantify the migration of pro-inflammatory monocytes towards adipose tissue specific media. This will then be compared to the other 3 groups to investigate the interaction between ethnicity, central obesity, and physical activity with the migration of pro-inflammatory monocytes.
  Metabolic markers will be analysed and presented in a participant characteristics table.
  Interventions: Behavioral: Habitual physical activity assessment

INTERVENTIONS:
Behavioral: Habitual physical activity assessment — 7 days habitual physical activity via accelerometry (ActiGraph GT3x). Specifically steps per day, light physical activity (minutes per day), and moderate to vigorous physical activity (minutes per day).

SUMMARY:
Being south Asian or centrally obese may be associated with an increased risk of inflammation. The investigators are seeking to investigate whether this is the case by recruiting white European and south Asian men who are lean or have central obesity. Further, the investigators wish to investigate whether physical activity influences the associations.

DETAILED DESCRIPTION:
Central obesity is associated with an increased risk of cardiovascular disease. Further, south Asians have been shown to be at an increased risk of cardiovascular disease compared to white Europeans.

Cardiovascular disease is underpinned by inflammation. Evidence suggests that people with obesity have a more pro-inflammatory and pro-migratory monocyte profile compared with individuals who are lean. The excessive monocyte migration contributes to metabolic dysfunction over time, increasing the risk of chronic disease. However, there is no evidence in south Asians.

One modifiable risk factor which may be able to influence this is physical inactivity, with higher levels of physical activity being associated with reduced inflammation. However, although south Asians are more at risk of cardiovascular disease than white Europeans, evidence suggests south Asians are also less physically active than white Europeans.

The investigators are looking to recruit south Asian and white European men who are lean or have central obesity to investigate 1) is there an association between ethnicity and the tethering and migration of pro-inflammatory monocytes? 2) is there an association between central obesity and the tethering and migration of pro-inflammatory monocytes, and is there an interaction with ethnicity? 3) do higher levels of physical activity influence the tethering and migration of pro-inflammatory monocytes, and is this influenced by ethnicity or central obesity?

To investigate this, the investigators are looking to recruit south Asian and white European men who are either centrally obese or lean. The investigators require 1 blood sample and the participants to wear an activity monitor for 7 days.

Peripheral blood mononuclear cells (PBMCs) will be isolated from the whole blood sample. Then, the investigators will quantify the migratory capacity of PBMCs to a fixed chemokine gradient over time. Further, the investigators will phenotype the monocytes to indicate the characteristics of the monocytes that migrate towards the chemokine mix.

The activity monitor will quantify habitual physical activity, which will be used in the statistical analyses to investigate whether physical activity may influence the response.

It is important to investigate as it will further scientific knowledge on the underpinnings of chronic disease and enable a better understanding on the role of physical activity to potentially reduce the risk.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers (including vaping)
* Not currently dieting

Exclusion Criteria:

* Musculoskeletal injury that has affected normal ambulation within the last month;
* Any muscle or bone injuries that influence physical activity
* Free from heart conditions and blood disorders
* Weight fluctuation greater than 3kg in the previous 3 months
* Taking anti-inflammatory medication

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants will be recruited from the local community using advertisements published online and across local facilities and shops.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Concentrations of classical monocytes. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as cells/uL.
Concentrations of intermediate monocytes. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as cells/uL.
Concentrations of non-classical monocytes. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as cells/uL.
Concentrations of CCR2+ monocytes. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as cells/uL.
Concentrations of CCR2+ classical monocytes. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as cells/uL.
Concentrations of CCR5+ monocytes. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as cells/uL.
Number of monocytes that migrated. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of classical monocytes that migrated. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of intermediate monocytes that migrated. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of non-classical monocytes that migrated. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of CCR2+ monocytes that migrated. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of CCR2+ classical monocytes that migrated. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of CCR5+ monocytes that migrated. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of monocytes that tethered. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of classical monocytes that tethered. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of intermediate monocytes that tethered. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of non-classical monocytes that tethered. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of CCR2+ monocytes that tethered. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of CCR2+ classical monocytes that tethered. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
Number of CCR5+ monocytes that tethered. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry. Presented as number of cells.
CCR2+ receptor expression. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry.
CCR5+ receptor expression. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via flow cytometry.

SECONDARY OUTCOMES:
Concentration of total cholesterol. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of total cholesterol. Presented as mmol/L.
Concentration of high-density lipoprotein cholesterol (HDL). | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of high-density lipoprotein cholesterol. Presented as mmol/L.
Concentration of low-density lipoprotein cholesterol (LDL). | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of low-density lipoprotein cholesterol. Presented as mmol/L.
Concentration of triacylglycerol. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of triacylglycerol. Presented as mmol/L.
Concentration of glucose. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of glucose. Presented as mmol/L.
Concentration of c-reactive protein. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of c-reactive protein. Presented as mg/L.
Concentration of interleukin-6. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of interleukin-6. Presented as pg/mL.
Concentration of non-esterified free fatty acids. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Fasted concentration of non-esterified free fatty acids. Presented as mmol/L.
Body fat percentage. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Body fat percentage determined via bioelectrical impedance analysis. Presented as percentage.
Lean mass. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Determined via bioelectrical impedance analysis. Presented in kilograms.
Waist circumference | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Waist circumference. Presented as centimetres.
Systolic blood pressure. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Presented as mmHg.
Diastolic blood pressure. | The outcome will be measured as a single-time point assessment in a fasted state on day 1.
  Presented as mmHg.
Light physical activity minutes per day. | Over 7 days +/- the assessment day
  Time spent participating in light physical activity. Presented as minutes per day.
Moderate-to-vigorous activity minutes per day. | Over 7 days +/- the assessment day
  Time spent participating in moderate-to-vigorous physical activity. Presented as minutes per day.
Daily steps. | Over 7 days +/- the assessment day
  Total daily steps. Presented as steps per day.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolette Bishop, Principal Investigator — Loughborough University
Locations (1):
- National Centre for Sport and Exercise Medicine, Loughborough, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data for all primary and secondary outcome measures will be made upon request.
Time Frame: The data will be available 6 months after publication for 12 months.
Access Criteria: Data will be available to other researchers who would like to run the same statistical methods we have used to check the interpretation of results.